CLINICAL TRIAL: NCT02486081
Title: Assistive Device Design, Development and Application-Smart Football for Movement Evaluation and Training in the Special Education Population
Brief Title: Development and Application-Smart Football for Movement Evaluation and Training in the Special Education Population
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 103-7262B
Record Dates: First submitted 2015-06-04; First posted 2015-07-01 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2018-01

CONDITIONS: Intellectual Disability
Keywords: Assistive device; the disabled; special education; movement analysis; system development
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- children with intelligent disabilities: children with ID will be measured via a smart soccer ball. Performance will be measured as acceleration, total time for completion, total distance
  Interventions: Device: smart soccer ball
- typical-developed children (TD): TD children will be measured via a smart soccer ball. Performance will be measured as acceleration, total time for completion, total distance
  Interventions: Device: smart soccer ball

INTERVENTIONS:
Device: smart soccer ball — smart soccer ball was used to measure participant's performance in total time and distance for completion, and acceleration

SUMMARY:
Children with disabilities are frequently ignored by the general population, hence the development of movement evaluation and training devices for use in special education settings are relatively overlooked. Usually the performance of these children is not stable and contains variations. Hence in order to get a complete picture of their sport performance, simply measuring movement time and distance is definitely not representative. With the rising attention from government regarding fitness and social participation of the disabled in recent years, developing a special-designed individual evaluation & training plan is of great importance. To achieve this goal, a device which is able to record the complete process of movement, and contains algorithm that can pick up the movement characteristics of children with disabilities is needed. The purpose of this study is to design and develop a smart soccer ball system for use in children with intellectual disabilities(ID), and to compare the performance between children with ID and the typically developed.

ELIGIBILITY:
Inclusion Criteria:

1. Intellectual disabilities (ID) group:

   * children with mild to moderate intellectual disabilities.
   * able to walk independently
   * can follow simple commands
2. Typical developed children:

   * age-matched TD children

Exclusion Criteria:

1. fracture or receive orthopedic surgery within six months.
2. Participate in regular soccer training.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children with intellectual disabilities
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
acceleration (in m/sec square) | one week
distance completed (in meters) | one week
time (in second) | one week

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National TaoYuan Special School, Taoyuan District
  - Chang Gung Univ., Taoyuan District